CLINICAL TRIAL: NCT00790049
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Day And Multiple Day Ascending Dose Study To Evaluate The Safety And Pharmacokinetics Of Orally Administered ARRY-371797 In Healthy Volunteers
Brief Title: A Safety Study of ARRY-371797 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ARRAY-797-107; C4411015 (Other: Pfizer)
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Healthy
MeSH Terms: interventions — ARRY-371797

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARRY-371797 (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral

INTERVENTIONS:
Drug: ARRY-371797, p38 inhibitor; oral — single dose and multiple dose, escalating
  Arms: ARRY-371797
Drug: Placebo; oral — matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 study, involving both 1-day and 8-day dosing periods, designed to test the safety of investigational study drug ARRY-371797 in healthy subjects. Approximately 48 healthy subjects from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or female between the ages of 18 and 60 years.
* Females must be of nonchildbearing potential.
* Body weight > 50 kg (110 lbs) and < 113 kg (250 lbs).
* Additional criteria exist.

Key Exclusion Criteria:

* A positive test for drugs or alcohol.
* Use of prescription or nonprescription drugs, herbal or dietary supplements, vitamins, or grapefruit juice within 14 days prior to first dose of study drug.
* Additional criteria exist.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10-31 (Actual); Primary Completion 2009-01-21 (Actual); Study Completion 2009-01-21 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, vital signs and electrocardiograms. | Duration of study
Characterize the pharmacokinetics (PK) of the study drug and a metabolite in terms of plasma concentrations. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.